CLINICAL TRIAL: NCT02547376
Title: Genetic and Telomere Characteristics of High of Grade Soft Tissue Sarcomas
Status: Terminated | Type: Observational
Why Stopped: Covid-19
Sponsor: University Hospitals, Leicester (Other)
Responsible Party: Sponsor
Other Study IDs: UHL 11353
Record Dates: First submitted 2015-03-18; First posted 2015-09-11 (Estimated); Last update posted 2020-10-14 (Actual); Status verified 2020-10

CONDITIONS: Soft Tissue Sarcoma
Keywords: Telomeres; Telomerase; Alternative lengthening of Telomeres Mechanism
MeSH Terms: conditions — Sarcoma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Soft tissue sarcoma tissue Blood (Plasma and Buffy coat) Saliva
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Eligible patients with Soft Tissue Sarcoma: Primary Soft Tissue Sarcoma group

SUMMARY:
Soft tissue sarcomas (STSs) are a rare group of cancers that can arise in any 'soft' tissue but commonly involve muscles, fat and nerves. Even following surgery and radiotherapy over 50% of tumours will recur or spread and at present, there is no reliable test that allows doctors to predict in which patients this will occur.

DNA that is not inside cells (cell-free or cfDNA) is present in very small quantities circulating in blood. In cancer patients some of this cfDNA comes from cancer cells. Analysis of cancer-derived cfDNA in patients with other cancers has shown that the quantity and characteristics of cfDNA changes with stage of disease and treatment. The researchers plan to investigate the abundance and persistence of cancer-derived cfDNA in STS patients at various stages of disease to investigate the potential role of these characteristics as biomarkers.

Selection of the genetic characters to be tracked in the patients' cfDNA is an important consideration. An established hallmark of a cancer cell is the ability to undergo an unlimited number of cell divisions. In normal human cells protective structures on the ends of chromosomes called telomeres provide a mechanism to limit the number of times a healthy cell can divide. This limitation has to be overcome in cancer cells for a tumour to form. This occurs by the activation of one of two telomere maintenance mechanisms (TMM) - either an enzyme called Telomerase or a mechanism known as Alternative Lengthening of Telomeres (ALT). In many sarcomas the activation of either TMM is associated with genetic changes (mutations) in a small number of genes. As these mutations are not present in normal cells but mark an essential feature of cancer cells (and their capacity for unlimited cell division) they are likely to be reliable markers of the presence of STS cells.

The investigators plan to develop sensitive, quantitative assays to detect TMM associated mutations in tumour derived cfDNA in the blood of patients with STSs, and track these mutations overtime. They will establish the amount of cancer-derived cfDNA in STS patients at the time of surgery, and persistence of this cfDNA during follow up visits following tumour resection and in the events of local tumour recurrence or spread (metastatic disease). Once these basic parameters are established analysis will be broadened to include other genes that are commonly mutated in STSs with a view of identifying other genetic characteristics that may also aid identification of patients at high risk of recurrence or spread. In summary all of the assays described above should facilitate better monitoring of patients with STS, and allow earlier treatment if STS recurs following surgery.

DETAILED DESCRIPTION:
Aims

The investigators plan a 2 year pilot observational study to:

* Identify and quantify circulating cell-fee DNA (cfDNA) in cases of Soft Tissue Sarcoma (STS)
* Investigate Telomere Maintenance Mechanisms (TMM) in STSs.
* Use TMM associated genetic mutations to identify and quantify tumour-derived cfDNA in STSs at time of tumour resection and throughout follow up
* Track the tumour derived cfDNA characteristics above over time and correlate with clinical outcome to identify potential STS biomarkers Hypotheses Based on findings in other cancers it is hypothesised that plasma cfDNA will be detectable in cases of STS. Given the key role telomere length maintenance plays in cancer cell development the investigators also hypothesise that TMM associated mutations will be present in tumour derived cfDNA, act as stable markers of STS tissue, and therefore increase in concentration as local recurrence or metastatic disease occurs.

Tumour derived cfDNA identification In months 0-3 sensitive assays to target known tumour-specific mutations will be developed. Using these on retrospectively collected tissues the investigators will verify that cfDNA can be detected (and quantified) in the plasma of patients with STSs.

Analysis of TMMs in STS tissue In months 3-12 tumour samples from every prospectively recruited sample will be analysed to establish which TMM is activated in STSs. Telomerase and ALT activity will each be assessed by published laboratory techniques.

Quantification and characterisation of TMM associated mutations / tumour derived cfDNA In months 10-12 quantitative Polymerase Chain Reaction based assays will be developed to identify the TMM associated mutations found to be most prevalent in STSs. In months 12-22 these assays will be used to identify and quantify these TMM associated mutations (and therefore also tumour-derived cfDNA) in the plasma samples taken from every prospectively recruited patient at time of surgery and throughout follow up.

Correlation of cfDNA characteristics with clinical outcome In months 22-24 cfDNA concentration, tumour-derived cfDNA concentration and the genetic characteristics of both will be correlated with clinical outcome measure including local recurrence, metastatic recurrence and death to determine these characteristics' potential as future biomarkers.

Patient recruitment / sample collection Patients will be recruited through the East Midlands Sarcoma Service. Samples already available will be collected from 2 sources to verify that cfDNA can be detected in STSs: Firstly 20 patients with metastatic disease will be asked to give consent for retrospective analysis of their tumour tissue already archived following histological analysis. One blood sample will also be collected from these patients for analysis. Secondly every STS sample already stored in the Nottingham Health Science Biobank, (Nottingham City Hospital) with an accompanying plasma sample also stored (15 at time of writing) will be analysed.

For the investigators remaining analysis between months 0-22 patients with non-metastatic high-grade STSs undergoing a planned resection locally will be approached to participate. 2013 figures suggest over 100 patients will be eligible for inclusion. Tumour tissue, blood, and unaffected muscle and saliva (2 sources of control DNA) will be collected at time of resection. Repeat blood samples will be collected 3 monthly until the end of recruitment.

ELIGIBILITY:
Inclusion Criteria:

1. Cases of nonmetastatic biopsy proven highgrade soft tissue sarcoma (STS) presenting to the East Midlands Sarcoma Service
2. Cases to be treated with curative intent with surgical resection (+/adjuvant therapy)

Exclusion Criteria:

1. Cases presenting with local or distant recurrence
2. Retroperitoneal soft tissue sarcomas
3. Patients unable to provide informed consent
4. Patients aged under 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient managed by East Midland Sarcoma Service with Soft Tissue Sarcoma undergoing attempted curative resection
Sampling Method: Non-Probability Sample
Enrollment: 77 (Actual)
Dates: Start 2015-02-12 (Actual); Primary Completion 2020-09-28 (Actual); Study Completion 2020-09-28 (Actual)

PRIMARY OUTCOMES:
Disease recurrence (local and distant) post surgery | 18 months

SECONDARY OUTCOMES:
Overall survival | 18 months

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospitals of Leicester NHS Trust, Leicester, Leicestershire, United Kingdom